CLINICAL TRIAL: NCT05717504
Title: STARGATE (Sweet spoT for cArdiac Rhythm monitorinG After sTrokE) Pilot Trial: A Pilot-feasibility Randomized Controlled Trial
Brief Title: Sweet spoT for cArdiac Rhythm monitorinG After sTrokE
Acronym: STARGATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 122103
Record Dates: First submitted 2023-01-13; First posted 2023-02-08 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Implantable Loop Recorder; Anticoagulant; Stroke; Atrial fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disclosure (Active Comparator): Group A (disclosure arm): patients and physicians will be informed about all AF episodes identified on ILR lasting for ≥6 minutes.
  Interventions: Device: Implantable Loop Recorder; Other: Quality of life survey
- Non-Disclosure (Active Comparator): Group B (non-disclosure arm): patients and physicians will be only informed about AF episodes identified on ILR lasting for ≥24h. This longer threshold is selected because of its association with increased risk of systemic embolism.
  Interventions: Device: Implantable Loop Recorder; Other: Quality of life survey

INTERVENTIONS:
Device: Implantable Loop Recorder — Patients will be implanted with a loop recorder. Patients will be given the choice of remove the loop recorder after the 12-months follow-up visit or at the end of its battery life (approximately 3 years)
Other: Quality of life survey — A quality of life survey will be performed at the end of the follow-up period. The survey will be done over the phone or in person if the follow-up visit is in person.

SUMMARY:
The goal of this clinical trial is to compare the use of long-term vs. shorter-term heart monitoring to detect atrial fibrillation after stroke.

Patients will be implanted with a loop recorder and will have study follow-up at 3-, 6- an 12-months after implantation.

The investigators will evaluate 24 patients, between the 3 centers, in the same way the investigators plan to evaluate a larger number of participants (>1000) in a future study. This will allow us to learn if such a study is possible, identify potential implementation challenges, and develop strategies to overcome those difficulties.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder. Its name comes from the fibrillation (i.e. quivering) of the two upper chambers (atria) of the heart instead of a coordinated contraction, causing a rapid, irregular heart rate. This irregular contraction is ineffective, leading to the development clots in the heart. These clots can travel through the bloodstream until they get stuck in a brain artery. Millions of brain cells that depend on the oxygen supplied by the blocked artery die within minutes. This is known as a stroke. Strong blood thinners known as anticoagulants can lower stroke risk by 64% in AF patients when the AF is detected on an electrocardiogram (ECG) or if it lasts more than 24h on a heart monitor. Therefore, doctors use cardiac monitors to record the heartbeats of stroke patients for up to 3 years. It was historically thought, but not proven, that if AF was found in stroke patients, using anticoagulants could prevent a second stroke. However, recent information suggests that using cardiac monitors in stroke patients increases AF detection and anticoagulants prescription without a reduction in the number of new strokes. The failure to prevent a second stroke is likely the consequence of cardiac monitors sometimes detecting very short-duration AFs, which may have a low risk of stroke. If AFs last only for a few minutes or hours, anticoagulants may not be needed.

Patients with a stroke and not know atrial fibrillation will be implanted with a loop recorder and randomized in two groups (disclosure arm and non-disclosure arm). Patients will have phone follow-up visits at 3, 6 and 12 months after implantation. A quality-of-life survey will be performed at the last study visit.

This study will assess if it is possible to organize a large clinical trial comparing the use of long-term vs. shorter-term heart monitoring. The investigators will evaluate 24 patients, between the 3 centers, in the same way, the investigators plan to evaluate a larger number of participants (>1000) in a future study. This will allow us to learn if such a study is possible, identify potential implementation challenges, and develop strategies to overcome those difficulties.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with cortical or subcortical, cryptogenic or non-cryptogenic acute ischemic stroke

Exclusion Criteria:

* AF on 24-h inpatient or Holter monitoring
* Atrial or ventricular thrombus
* Other major-risk cardioembolic sources (e.g., mechanical valve)
* Other indications (e.g., venous thromboembolism) or contraindications for OACs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled at in 6 months | 6 months
  Median and interquartile range recruitment rate. We will use this rate to estimate the number of sites and enrollment duration required for a larger RCT.

SECONDARY OUTCOMES:
Screened, declined and dropouts. | 2 years
  1. proportion and 95% confidence intervals (95% CI) of stroke patients needed to screen per patient invited to participate
  2. proportion and 95% CI of patients declining participation
  3. proportion and 95% CI of dropouts at the end of follow-up.
Number of clinical endpoint events per diagnostic arm | 2 years
  The investigators will apply standard descriptive statistics to report the number of clinical endpoint events per diagnostic arm. The primary composite efficacy endpoint to be used in larger RCT is stroke recurrence (ischemic or hemorrhagic), systemic embolism, MACE (myocardial infarction and admission for decompensated AF or heart failure), and death. The primary safety endpoint will be major bleeding (ISTH definition).These data and results from prior studies will be used to estimate the final sample size and required number of sites for the larger RCT.
Quality of life survey analysis | 2 years
  The investigators will perform a qualitative and quantitative analysis of the results of the ILR-specific quality of life survey. The analysis will be reviewed by the team and PWLE. We will use this information to improve patients' experiences in a larger RCT
AF timing of diagnosis | 2 years
  The investigators will evaluate different measures of AF timing of diagnosis :Time to first AF diagnosis (DD:HH)
AF burden (1) | 2 years
  The investigators will evaluate different measures of AF burden:
  Total AF burden at 3, 6, and 12 months post-ILR insertion (sum of the duration of all AF episodes, HH:MM:SS).
  Characterizing these measures will allow us to choose the best AF burden definition for a larger RCT.
AF burden (2) | 2 years
  The investigators will evaluate different measures of AF burden:
  Maximum duration of the longest AF episode. Characterizing these measures will allow us to choose the best AF burden definition for a larger RCT.
AF burden (3) | 2 years
  The investigators will evaluate different measures of AF burden:
  Relative AF burden (total AF burden/net monitoring time), (4) AF Pattern (number of AF episodes and time of occurrence), (5) Other ECG monitoring findings (premature atrial complexes, interatrial block, etc.). Characterizing these measures will allow us to choose the best AF burden definition for a larger RCT.
AF burden (4) | 2 years
  The investigators will evaluate different measures of AF burden:
  AF Pattern (number of AF episodes and time of occurrence). Characterizing these measures will allow us to choose the best AF burden definition for a larger RCT.
AF burden (5) | 2 years
  The investigators will evaluate different measures of AF burden:
  Other ECG monitoring findings (premature atrial complexes, interatrial block, etc.). Characterizing these measures will allow us to choose the best AF burden definition for a larger RCT.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano A Sposato, MD, MBA, Principal Investigator — LHSC - Western University